CLINICAL TRIAL: NCT02006654
Title: Randomised, Double-blind, Parallel-group, Placebo-controlled Study of Idalopirdine in Patients With Mild - Moderate Alzheimer's Disease Treated With an Acetylcholinesterase Inhibitor
Brief Title: Study of Idalopirdine in Patients With Mild - Moderate Alzheimer's Disease Treated With an Acetylcholinesterase Inhibitor
Acronym: STARBRIGHT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14863A; 2012-004765-40 (EudraCT Number)
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — (2-(6-fluoro-1H-indol-3-yl)-ethyl)-(3-(2,2,3,3-tetrafluoropropoxy)benzyl)amine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo adjunct to base treatment with an AChEI
  Interventions: Drug: Placebo
- Idalopirdine 60 mg (or 30 mg) (Experimental): Idalopirdine adjunct to base treatment with an AChEI
  Interventions: Drug: Idalopirdine

INTERVENTIONS:
Drug: Placebo — Once daily, matching placebo capsules, orally
  Arms: Placebo
Drug: Idalopirdine — Once daily, encapsulated tablets, orally
  Other Names: Lu AE58054
  Arms: Idalopirdine 60 mg (or 30 mg)

SUMMARY:
To establish efficacy of idalopirdine as adjunctive therapy to acetylcholinesterase inhibitors (AChEIs) for symptomatic treatment of patients with mild-moderate Alzheimer's disease (AD).

DETAILED DESCRIPTION:
The study consisted of a screening period (up to 2-week period from screening to randomization), a 24-week double-blind treatment period with placebo or idalopirdine 60mg/day as adjunctive therapy to an acetylcholinesterase inhibitor (donepezil 10mg/day, rivastigmine at the patient's individual maintenance dose, or galantamine at the patient's individual maintenance dose), and a 4-week safety follow-up period following study completion or withdrawal from treatment. The dose could be decreased once during the study to 30mg/day if 60mg/day was not well tolerated in the opinion of the investigator. The dose could be increased again to 60mg/day, after which the dose was kept fixed for the remainder of the study. Dose changes were permitted until Week 12 (Visit 5).

ELIGIBILITY:
Inclusion Criteria:

* The patient has a knowledgeable and reliable caregiver.
* The patient is an outpatient.
* The patient has probable AD.
* The patient has mild to moderate AD.
* Stable treatment with an AChEI.
* The patient, if a woman, must have had her last natural menstruation ≥24 months prior to baseline, OR be surgically sterile.
* The patient, if a man, agrees to protocol-defined use of effective contraception if his female partner is of childbearing potential, OR must have been surgically sterilised prior to the screening visit.

Exclusion Criteria:

* The patient has evidence of any clinically significant neurodegenerative disease, or other serious neurological disorders other than AD.
* The patient has a Diagnostic and Statistical Manual of Mental Disorders, 4th edition, Text Revision (DSM-IV-TR) Axis I disorder other than AD.
* The patient has evidence of clinically significant disease.
* The patient's current AChEI therapy is likely to be interrupted or discontinued during the study.
* The patient is currently receiving memantine or has taken memantine within 2 months prior to screening.

Other inclusion and exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 734 (Actual)
Dates: Start 2014-03; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (107):
- United States (26):
  - US612, Mesa, Arizona
  - US625, Bellflower, California
  - US626, Costa Mesa, California
  - US604, Oxnard, California
  - US627, Santa Ana, California
  - US609, Danbury, Connecticut
  - US614, Norwalk, Connecticut
  - US608, Deerfield Beach, Florida
  - US616, Hialeah, Florida
  - US620, Miami, Florida
  - US603, North Palm Beach, Florida
  - US631, Port Charlotte, Florida
  - US622, Elk Grove Village, Illinois
  - US611, Elkhart, Indiana
  - US606, Prairie Village, Kansas
  - US601, Farmington Hills, Michigan
  - US607, St Louis, Missouri
  - US613, Lawrenceville, New Jersey
  - US635, Paterson, New Jersey
  - US630, Toms River, New Jersey
  - US621, Albany, New York
  - US632, Staten Island, New York
  - US633, Charlotte, North Carolina
  - US623, Oklahoma City, Oklahoma
  - US618, Norristown, Pennsylvania
  - US619, Houston, Texas
- Australia (7):
  - AU603, Caulfield
  - AU609, Glen Iris
  - AU602, Heidelberg West
  - AU604, Kanwal
  - AU606, Newcastle
  - AU601, West Perth
  - AU610, Woodville South
- Brazil (3):
  - BR608, Belo Horizonte
  - BR609, Itapira
  - BR607, Rio de Janeiro
- Czechia (8):
  - CZ602, Choceň
  - CZ608, Choceň
  - CZ605, Havlíčkův Brod
  - CZ606, Kladno
  - CZ603, Pilsen
  - CZ601, Prague
  - CZ604, Prague
  - CZ607, Praha 10 - Strasnice
- Germany (14):
  - DE612, Bad Homburg
  - DE610, Bad Honnef
  - DE609, Berlin
  - DE617, Berlin
  - DE604, Erbach im Odenwald
  - DE611, Freiburg im Breisgau
  - DE607, Gelsenkirchen
  - DE605, Homburg
  - DE608, Karlstadt am Main
  - DE602, Mittweida
  - DE601, Munich
  - DE606, Rostock
  - DE603, Ulm
  - DE616, Unterhaching
- Israel (5):
  - IL605, Bat Yam
  - IL601, Haifa
  - IL604, Holon
  - IL602, Ramat Gan
  - IL603, Tel Aviv
- Mexico (6):
  - MX602, México
  - MX601, Monterrey
  - MX603, Monterrey
  - MX604, Monterrey
  - MX605, Monterrey
  - MX606, Saltillo
- Serbia (3):
  - RS602, Belgrade
  - RS603, Kragujevac
  - RS601, Novi Sad
- Singapore (2):
  - SG601, Singapore
  - SG602, Singapore
- Slovakia (5):
  - SK601, Banská Bystrica
  - SK603, Bratislava
  - SK605, Bratislava
  - SK604, Rimavská Sobota
  - SK602, Svidník
- South Korea (4):
  - KR601, Seongnam-si
  - KR602, Seoul
  - KR603, Seoul
  - KR604, Seoul
- Spain (12):
  - ES601, Barcelona
  - ES603, Barcelona
  - ES604, Barcelona
  - ES608, Barcelona
  - ES611, Bilbao
  - ES612, Burgos
  - ES602, Lleida
  - ES613, Madrid
  - ES610, Sant Cugat del Vallès
  - ES606, Seville
  - ES605, Terrassa
  - ES607, Valencia
- Switzerland (4):
  - CH603, Biel
  - CH605, Lausanne
  - CH602, Les Acacias
  - CH601, Schlieren
- Turkey (Türkiye) (6):
  - TR602, Balova
  - TR601, Istanbul
  - TR603, Istanbul
  - TR605, Istanbul
  - TR606, Izmir
  - TR607, Samsun
- United Kingdom (2):
  - GB601, Brentford
  - GB603, Northampton

REFERENCES:
- [Derived] Ballard C, Atri A, Boneva N, Cummings JL, Frolich L, Molinuevo JL, Tariot PN, Raket LL. Enrichment factors for clinical trials in mild-to-moderate Alzheimer's disease. Alzheimers Dement (N Y). 2019 May 20;5:164-174. doi: 10.1016/j.trci.2019.04.001. eCollection 2019. PMID 31193334
- [Derived] Cummings JL, Atri A, Ballard C, Boneva N, Frolich L, Molinuevo JL, Raket LL, Tariot PN. Insights into globalization: comparison of patient characteristics and disease progression among geographic regions in a multinational Alzheimer's disease clinical program. Alzheimers Res Ther. 2018 Nov 24;10(1):116. doi: 10.1186/s13195-018-0443-2. PMID 30474567
- [Derived] Atri A, Frolich L, Ballard C, Tariot PN, Molinuevo JL, Boneva N, Windfeld K, Raket LL, Cummings JL. Effect of Idalopirdine as Adjunct to Cholinesterase Inhibitors on Change in Cognition in Patients With Alzheimer Disease: Three Randomized Clinical Trials. JAMA. 2018 Jan 9;319(2):130-142. doi: 10.1001/jama.2017.20373. PMID 29318278

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Idalopirdine 60 mg (or 30 mg)
Started | 369 | 365
Treated | 365 | 363
Completed | 324 | 321
Not Completed | 45 | 44
Not completed — Withdrawal before treatment | 4 | 2
Not completed — Adverse Event | 16 | 17
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 14 | 12
Not completed — Protocol Violation | 5 | 8
Not completed — Lost to Follow-up | 1 | 0
Not completed — patient's will | 2 | 1
Not completed — insufficient compliance | 1 | 0
Not completed — worsening cognitive condition | 0 | 1
Not completed — faecal incontinence | 0 | 1
Not completed — mood disorder | 0 | 1
Not completed — disallowed medication | 1 | 0
Not completed — moving out of state | 0 | 1

BASELINE CHARACTERISTICS:
Population: A total of 734 patients were randomized into the study but 6 patients were not treated (did not receive IMP). The baseline analysis population only consist of patients who have been treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Idalopirdine 60 mg (or 30 mg) | Total
Number analyzed (Participants) | 365 | 363 | 728
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.2 (8.0) | 73.6 (8.6) | 73.9 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 135 | 266
  Male | 234 | 228 | 462
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 14
  Not Hispanic or Latino | 33 | 33 | 66
  Unknown or Not Reported | 324 | 324 | 648
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | NA — Information has not been collected | NA — Information has not been collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Asian | 40 | 39 | 79
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 7 | 19
  White | 292 | 299 | 591
  More than one race | NA — Information has not been collected | NA — Information has not been collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 21 | 18 | 39
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 17 | 15 | 32
  United States | 41 | 39 | 80
  Czechia | 42 | 37 | 79
  United Kingdom | 7 | 4 | 11
  Switzerland | 2 | 2 | 4
  Spain | 65 | 62 | 127
  South Korea | 19 | 20 | 39
  Turkey | 15 | 14 | 29
  Brazil | 23 | 21 | 44
  Mexico | 25 | 23 | 48
  Slovakia | 27 | 29 | 56
  Israel | 7 | 9 | 16
  Australia | 19 | 23 | 42
  Germany | 37 | 43 | 80
  France | 9 | 11 | 20
MMSE total score at screening [Mean (Standard Deviation); unit: units on a scale] — Measure Description: The Mini Mental State Examination (MMSE) is an 11-item test to assess the cognitive aspects of mental function. The subtests assess orientation, memory, attention, language, and visual construction. The scores for each item is dichotomous (1 = response is correct, 0 = response is incorrect). Total score of the 11 items ranges from 0 to 30 (higher score indicates lower deficit).
  units on a scale | 17.5 (3.0) | 17.2 (2.9) | 17.3 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognition
Description: Change from baseline to Week 24 in Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog) total score.
  The Alzheimer's Disease Assessment Scale - Cognitive subscale (ADAS-cog) is a 11-item neuropsychological test that assess the severity of cognitive impairment. The items determine the patient's orientation, memory, language, and praxis. Total score of the 11 items range from 0 to 70 (lower score indicates lower cognitive impairment).
Time Frame: Baseline and Week 24
Population: All patients who took at least one dose of placebo or idalopirdine, and who had a valid baseline assessment and at least one valid post-baseline assessment of the primary outcome measure in the 24-week treatment period (Full-analysis Set). For secondary outcome measures, the number of participants who had the respective outcome measure assessed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Idalopirdine 60 mg (or 30 mg)
Number analyzed (Participants) | 356 | 361
units on a scale | 0.68 (0.37) | 0.13 (0.38)
Statistical Analysis 1: Comparison: Placebo vs Idalopirdine 60 mg (or 30 mg); For demonstrating efficacy, change in cognition (ADAS-cog) and either change in daily functioning (ADCS-ADL23) or change in global clinical impression (ADCS-CGIC) had to show statistically significant favourable differences compared to placebo at Week 24. Multiple testing procedures were used to control the overall type 1 error at 5%. The null hypothesis of no difference in mean change from baseline in ADAS-cog total score at Week 24 was tested for idalopirdine at significance level 5%; Test type: Superiority; p = 0.2365, Mixed Models Analysis — Corrected for multiplicity; Adjusted for effects of country, MMSE stratum-by-week, treatment-by-week, base treatment stratum-by-week, and baseline score-by-week interactions; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-1.45 to 0.36], Standard Error of Mean 0.46 — A negative mean difference indicates a treatment effect in favor of idalopirdine

2. Secondary Outcome: Change in Global Impression
Description: Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (ADCS-CGIC) score at Week 24.
  The Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change is a semi-structured interview to assess clinically relevant changes in patients with AD. The items determine cognition, behavior, social and daily functioning. Severity at baseline is rated on a 7-point scale from 1 (normal, not ill at all) to 7 (among the most extremely ill patients). The clinically relevant change from baseline is rated on a 7-point scale from 1 (marked improvement) to 7 (marked worsening).
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Idalopirdine 60 mg (or 30 mg)
Number analyzed (Participants) | 353 | 357
units on a scale | 4.32 (0.07) | 4.39 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Idalopirdine 60 mg (or 30 mg); For demonstrating efficacy, change in cognition (ADAS-cog) and either change in daily functioning (ADCS-ADL23) or change in global clinical impression (ADCS-CGIC) had to show statistically significant favourable differences compared to placebo at Week 24. Multiple testing procedures were used to control the overall type 1 error at 5%. The null hypothesis of no difference in mean change from baseline in ADAS-cog total score at Week 24 was tested at significance level 5%; Test type: Superiority; p = 0.4064, Mixed Models Analysis — Corrected for multiplicity according to the multiple testing procedure; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.09 to 0.23], Standard Error of Mean 0.08 — A negative mean difference indicates a treatment effect in favor of idalopirdine

3. Secondary Outcome: Change in Daily Functioning
Description: Change from baseline to Week 24 in Alzheimer's Disease Cooperative Study - Activities of Daily Living Inventory (ADCS-ADL23) total score.
  The Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL23) is a 23-item clinician-rated inventory to assess activities of daily living (conducted with a caregiver or informant). Each item comprises a series of hierarchical sub-questions, ranging from the highest level of independent performance to a complete loss for each activity. Total score of the 23 items ranges from 0 to 78 (higher score indicates lower disability).
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Idalopirdine 60 mg (or 30 mg)
Number analyzed (Participants) | 356 | 361
units on a scale | -1.72 (0.50) | -1.05 (0.51)
Statistical Analysis 1: Comparison: Placebo vs Idalopirdine 60 mg (or 30 mg); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.4064, Mixed Models Analysis — Corrected for multiplicity according to the multiple testing procedure; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.67, 95% CI 2-sided [-0.57 to 1.92], Standard Error of Mean 0.63 — A positive mean difference indicates a treatment effect in favour of idalopirdine

4. Secondary Outcome: Change in Behavioural Disturbance
Description: Change from baseline to Week 24 in Neuropsychiatric Inventory (NPI) total score
  The Neuropsychiatric Inventory is a 12-item structured interview with a caregiver to assess behavioural disturbances. The NPI comprises 10 behavioural and 2 neurovegetative items. Each item consists of a screening question and several sub-questions that are rated no (not present) or yes (present). Each item is then rated for frequency (a 4-point scale from 1 [occasionally] to 4 [very frequent]) and severity (a 3-point scale from 1 [mild] to 3 [marked]). The total NPI score is the frequency ratings multiplied by the severity ratings and ranges from 0 to 144 (higher score indicates worse outcome).
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Idalopirdine 60 mg (or 30 mg)
Number analyzed (Participants) | 356 | 361
units on a scale | -0.46 (0.53) | -0.74 (0.54)

5. Secondary Outcome: Change in Individual Behavioural Disturbance Items
Description: Change in single NPI item scores at Week 24.
  The Neuropsychiatric Inventory is a 12-item structured interview with a caregiver to assess behavioural disturbances. The NPI comprises 10 behavioural and 2 neurovegetative items. Each item consists of a screening question and several sub-questions that are rated no (not present) or yes (present). Each item is then rated for frequency (a 4-point scale from 1 [occasionally] to 4 [very frequent]) and severity (a 3-point scale from 1 [mild] to 3 [marked]). Total score for each single NPI item ranges from 0-12 (frequency multiplied by severity), where higher scores represent worse outcome.
Time Frame: Baseline and Week 24
Population: All patients who took at least one dose of placebo or idalopirdine and who had a valid baseline assessment and at least one valid post-baseline assessment of the primary outcome measure in the 24-week treatment period (Full-analysis Set). For secondary outcome measures, the number of participants who had the respective outcome measure/item assessed
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Idalopirdine 60 mg (or 30 mg)
Number analyzed (Participants) | 356 | 361
units on a scale
  Delusions | -0.00 (0.10) | 0.03 (0.10)
  Hallucinations | 0.05 (0.06) | 0.08 (0.06)
  Agitation/aggression | 0.15 (0.11) | 0.03 (0.11)
  Depression/dysphoria | -0.28 (0.09) | -0.18 (0.09)
  Anxiety | -0.16 (0.09) | -0.07 (0.09)
  Elation/euphoria | 0.02 (0.04) | 0.03 (0.04)
  Apathy/indifference | -0.06 (0.15) | -0.19 (0.15)
  Disinhibition | 0.12 (0.08) | -0.00 (0.08)
  Irritability/lability | 0.10 (0.12) | -0.04 (0.12)
  Aberrant motor behaviour | 0.08 (0.11) | 0.11 (0.11)
  Sleep | -0.13 (0.11) | -0.12 (0.11)
  Appetite/eating disorder | -0.25 (0.12) | -0.21 (0.12)

6. Secondary Outcome: Change in NPI Anxiety Item Score in Patients With an NPI Anxiety Item Score of at Least 2 at Baseline
Description: Change from baseline to Week 24 in NPI anxiety item score in patients with an NPI anxiety item score of at least 2 at baseline
  The Neuropsychiatric Inventory is a 12-item structured interview with a caregiver to assess behavioural disturbances. The NPI comprises 10 behavioural and 2 neurovegetative items. Each item consists of a screening question and several sub-questions that are rated no (not present) or yes (present). Each item is then rated for frequency (a 4-point scale from 1 [occasionally] to 4 [very frequent]) and severity (a 3-point scale from 1 [mild] to 3 [marked]). The total score for the NPI anxiety item ranges from 0-12 (frequency multiplied by severity), where a higher score represents a worse outcome.
Time Frame: Baseline and Week 24
Population: All patients who took at least one dose of placebo or idalopirdine and who had a valid baseline assessment and at least one valid post-baseline assessment of the primary outcome measure in the 24-week treatment period (Full-analysis Set). For secondary outcome measures, the number of participants who had the respective outcome/item measure assessed
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Idalopirdine 60 mg (or 30 mg)
Number analyzed (Participants) | 86 | 83
units on a scale | -1.93 (0.32) | -1.52 (0.33)

7. Secondary Outcome: Clinical Improvement
Description: Clinical response at Week 24 (based on pre-specified ADAS-cog, ADCS-ADL23, and ADCS-CGIC changes [change in ADAS-cog below or equal to -4, change in ADCS-ADL23 at least 0, and ADCS-CGIC below or equal to 4])
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Idalopirdine 60 mg (or 30 mg)
Number analyzed (Participants) | 324 | 321
Participants | 32 | 35

8. Secondary Outcome: Clinical Worsening
Description: Clinical worsening at Week 24 (Based on pre-specified ADAS-cog, ADCS-ADL23, and ADCS-CGIC changes [change in ADAS-cog above or equal to 4, change in ADCS-ADL23 below 0, and ADCS-CGIC above 4])
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Idalopirdine 60 mg (or 30 mg)
Number analyzed (Participants) | 324 | 321
Participants | 37 | 40

9. Secondary Outcome: Change in Cognitive Aspects of Mental Function
Description: Change from baseline to Week 24 in Mini Mental State Examination (MMSE).
  The Mini Mental State Examination (MMSE) is an 11-item test to assess the cognitive aspects of mental function. The subtests assess orientation, memory, attention, language, and visual construction. The scores for each item is dichotomous (1 = response is correct, 0 = response is incorrect). Total score of the 11 items ranges from 0 to 30 (higher score indicates lower deficit).
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Idalopirdine 60 mg (or 30 mg)
Number analyzed (Participants) | 323 | 320
units on a scale | -0.64 (0.20) | -0.35 (0.20)

10. Secondary Outcome: Change in Health-related Quality of Life (EQ-5D) Utility Score
Description: Change from baseline to Week 24 in EuroQol 5-dimensional (EQ-5D) utility score
  The EQ-5D is a patient-reported assessment that measures the patient's well-being. It consists of an utility score based on 5 descriptive items (mobility, self-care, usual activities, pain/discomfort, and depression/anxiety) and a Visual Analogue Scale (VAS). Each descriptive item is rated on a 3-point index ranging from 1 (no problems) to 3 (extreme problems) that is used for calculating a single summary index (from 0 to 1). A higher EQ-5D score indicates a worse outcome.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Idalopirdine 60 mg (or 30 mg)
Number analyzed (Participants) | 351 | 354
units on a scale | -0.01 (0.01) | -0.00 (0.01)

11. Secondary Outcome: Change in Health-related Quality of Life (EQ-5D VAS)
Description: Change from baseline to Week 24 in EQ-5D Visual Analogue Scale (EQ-5D VAS).
  The EQ-5D is a patient-reported assessment that measures the patient's well-being. It consists of an utility score based on 5 descriptive items (mobility, self-care, usual activities, pain/discomfort, and depression/anxiety) and a Visual Analogue Scale (VAS). The VAS ranges from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Idalopirdine 60 mg (or 30 mg)
Number analyzed (Participants) | 351 | 353
units on a scale | -0.40 (1.00) | 0.51 (1.02)

ADVERSE EVENTS:
Time Frame: Baseline to end of study
Description: Treatment-Emergent Adverse Events are reported in this section
Groups:
- Idalopirdine 60 mg: Idalopirdine adjunct to base treatment with an AChEI
  Idalopirdine: Once daily, encapsulated tablets, orally
Arm/Group | Placebo | Idalopirdine 60 mg
All-Cause Mortality (participants affected / at risk) | 1/365 | 0/363
Serious Adverse Events (participants affected / at risk) | 22/365 | 28/363
Other Adverse Events (participants affected / at risk) | 64/365 | 82/363
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=365) | Idalopirdine 60 mg (N=363)
Bradycardia (Cardiac disorders) | 0 | 2
Left ventricular failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 1
Retinal detachment (Eye disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 1 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 5
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 2 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Electrocardiogram st segment depression (Investigations) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/234 | 1/228
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haematoma (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Intracranial haematoma (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Agitation (Psychiatric disorders) | 1 | 0
Behavioural and psychiatric symptoms of dementia (Psychiatric disorders) | 0 | 1
Personality disorder (Psychiatric disorders) | 1 | 0
Azotaemia (Renal and urinary disorders) | 1 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Hypertensive emergency (Vascular disorders) | 0 | 1
Internal haemorrhage (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Peripheral venous disease (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=365) | Idalopirdine 60 mg (N=363)
Accidental overdose (Injury, poisoning and procedural complications) | 43 | 40
Fall (Injury, poisoning and procedural complications) | 21 | 19
Aspartate aminotransferase increased (Investigations) | 3 | 19
Gamma-glutamyltransferase increased (Investigations) | 2 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No